CLINICAL TRIAL: NCT05135338
Title: Comparison Between a Senior and a Junior Interpretation of a Chest X-ray in the Diagnosis of Heart Failure
Brief Title: Chest X-ray in Diagnosis of Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, chief of the Emergency departement in CHU fattouma Bourguiba Monastir , PhD, University of Monastir
Other Study IDs: Chest-X-ray/HF
Record Dates: First submitted 2021-11-18; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Chest X-ray ; Heart Failure
Keywords: chest x-ray; heart failure; diagnosis; senior; non-senior
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- answer 1: a senior emergency physician on interpretation of chest x-ray and blinded to the final diagnosis .
- answer 2: a resident or an intern interpretation of chest x-ray and blinded to the final diagnosis

SUMMARY:
The objective of this study is to compare the performance of x-chest ray in the diagnosis of acute cardiac insuficiency through the interpretation of a senior and a non-senior.

DETAILED DESCRIPTION:
Acute cardiac insufficiency (ICA) is a leading cause of acute dyspnea in the emergency department (SU) and is associated with a higher risk of morbidity and mortality.

An increasing number of tools for better ICA diagnosis are available in the SUs. However, there is likely room to improve the ICA diagnostic approach using widely available routine tools, including chest x-ray .

Chest x-ray is a rapid and inexpensive method that is routinely performed in an emergency in patients with acute dyspnea. This is the first-line diagnostic imaging modality recommended in the guidelines.

The objective of this study is to compare the performance of x-chest ray in the diagnosis of acute cardiac insuficiency through the interpretation of a senior and a non-senior.

A senior emergency physician or resident and an intern, perform a reading of chest x-ray in any included patient by answering to following questions:

Is there cardiomegaly? Calculation of the cardio-thoracic index Is there a vascular distribution towards the vertices, if so is it uni or bilateral? Is there pleurisy, if so is it uni or bilateral? Is there an interstitial syndrome, if so is it uni or bilateral? Is there an alveolar syndrome, if so if so is it single or bilateral? Is the diagnosis of heart failure very likely, likely or unlikely? Then there will be a comparison of the two answers.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 All dyspnea acute non-traumatic A resident or intern in medicine and a senior are available to read chest x-ray within 24 hours of admission

Exclusion Criteria:

* Age under 18
* Post traumatic dyspnea
* Patient not requiring hospitalization
* Mechanical ventilation from the start
* Cardio-respiratory arrest
* Pregnant woman
* And any patient who cannot achieve reproducibility within 24 hours of admission.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: alla patients admitted to th ED with acurte dyspnea who have recieved chest x- ray .
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
The reproductibility of chest x-ray in the diagnosis of heart failure | 0 days
  Comparison of the two answers of a senior and non -senior emergency physician chest x- ray interpretation in the probability of heart failure diagnosis .

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, PhD, Principal Investigator — University of Monastir
Locations (1):
- Fattouma Bourguiba Monastir University Hospital Center, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided